CLINICAL TRIAL: NCT03077776
Title: Tracking Triple-negative Breast Cancer Evolution Through Therapy
Acronym: TRACERX-TNBC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UC-0105/1614; ID RCB: 2016-A01177-44 (Other: ANSM)
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Triple-Negative Breast Neoplasm
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All included patients (Experimental): Patients will undergo a biopsy and provide a blood sample prior to initiating standard neoadjuvant chemotherapy. Additional tissue samples will be collected at the following time points:
  1. (optional) biopsy of primary tumour after 4 cycles of neoadjuvant chemotherapy
  2. At the time of surgery (samples of the primary tumour and lymph nodes which are surplus to diagnostic requirements).
  3. Biopsy of a metastatic site in the event of disease recurrence.
  Blood samples will be obtained during neoadjuvant chemotherapy, prior to surgery and at 6-month intervals for up to 5 years post-surgery. In the event of recurrent disease, blood samples will be collected i) at the time of recurrence, ii) at the first CT scan on treatment and iii) at each subsequent relapse for up to 5 years post-surgery.
  Interventions: Procedure: Biopsy; Procedure: Biopsy (optional); Procedure: Biopsy (metastatic)

INTERVENTIONS:
Procedure: Biopsy — Biopsy of primary tumour to be performed prior to initiation of neoadjuvant chemotherapy
Procedure: Biopsy (optional) — [Optional] biopsy of primary tumour to be performed after 4 weeks of neoadjuvant chemotherapy
Procedure: Biopsy (metastatic) — Biopsy of metastatic site to be performed at the time of relapse

SUMMARY:
A prospective multicentre study which aims to examine the relationship between intratumour heterogeneity (ITH) and pathological response to neoadjuvant chemotherapy in patients with histological confirmation of triple-negative breast cancer (TNBC) who are eligible for neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-years or older
2. Patients with histological confirmation of invasive breast cancer with known receptor status suitable for neoadjuvant chemotherapy as assessed by the local investigator
3. Estrogen receptor (ER)- and progesterone receptor (PR)-negative as defined by ≤1% of positive staining on immunohistochemistry
4. Human epidermal growth factor receptor 2 (HER2)-negative as defined by American Society of Clinical Oncology / College of American Pathologists guidelines
5. T1c-4 tumours (including inflammatory cancers), with any nodal status non candidate for conservative surgery upfront. Bilateral or multifocal cancer is permitted provided that all sites are HER2-negative and at least one site is ER- and PR-negative.
6. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses
7. Patient with social insurance coverage

Exclusion Criteria:

1. Confirmed metastatic disease at initial presentation
2. Any contraindication to the biopsy procedure
3. Previous or current malignancies of other origin within the last 5 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin
4. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
5. Individuals deprived of liberty or placed under the authority of a tutor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete response (pCR) | pCR will be defined at the time of surgery on the tumor specimen
  pCR is defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled ipsilateral lymph nodes (i.e., ypT0/Tis ypN0 in the current American Joint Committee on Cancer [AJCC] staging system)

SECONDARY OUTCOMES:
Invasive disease-free survival | from surgery until 5 years post-surgery
  the time from neoadjuvant treatment initiation until the date of the first occurrence of one of the following events: invasive ipsilateral breast tumour recurrence (same breast), local /regional invasive recurrence, invasive contra lateral breast cancer, appearance of metastasis, second primary invasive cancer (non-breast cancer), ipsilateral ductal carcinoma in situ, contralateral ductal carcinoma in situ, death attributable to any cause.
Overall survival | from surgery until 5 years post-surgery
  the time from neoadjuvant treatment until death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Monica ARNEDOS, MD, Principal Investigator — Gustave Roussy Cancer Campus
Locations (10):
- France (10):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Centre Leon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancerologie de l'Ouest, Nantes
  - Centre Eugène Marquis, Rennes
  - Centre Paul Strauss, Strasbourg
  - Hopitaux universitaire de strasbourg - Hopital civil, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNICANCER official website — http://www.unicancer.fr/